CLINICAL TRIAL: NCT02794012
Title: Periodontal Inflammation and Immunity in Preclinical Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Rheumatology Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 15-2288
Record Dates: First submitted 2016-05-26; First posted 2016-06-08 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Rheumatoid Arthritis; Periodontal Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- At-Risk Rheumatoid Arthritis subjects
- Early Rheumatoid Arthritis subjects
- Healthy Controls
- Non-Rheumatoid Arthritis Autoimmune Controls

SUMMARY:
The purpose of this study is to evaluate the association of Rheumatoid Arthritis (RA)-related antibodies and periodontal inflammation in subjects at-risk for Rheumatoid Arthritis. Subjects will undergo periodontal and joint examinations, as well as collection of body fluids to measure Rheumatoid Arthritis-related antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis-antibody positivity (anti-CCP) in the absence of arthritis or
* Early RA <36 months since diagnosis

Exclusion Criteria:

* Pregnancy
* Antibiotic use prior to dental procedures or cleanings
* Wear dentures
* <18 years old

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include: subjects at-risk for RA, subjects with early RA, and healthy controls >40 years old.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Degree of periodontal disease by oral examinations according to the American Academy of Periodontology (AAP) guidelines | 1 day

SECONDARY OUTCOMES:
Frequency of bacterial communities of the periodontium by bacterial diversity (e.g. Shannon Diversity Index) and bacterial load (qPCR) | 1 day
Frequency of Rheumatoid Arthritis-related antibodies in blood and mucosal sites using Rheumatoid Factor and Anti-Citrullinated Protein Antibody assays | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay B Kelmenson, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Barbara Davis Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No